CLINICAL TRIAL: NCT01398111
Title: Open-label, Randomized, Single-dose, Placebo-controlled, 4-way Crossover Study to Investigate the Pharmacokinetic Interaction of Glycopyrrolate and Formoterol in Healthy Subjects.
Brief Title: Pharmacokinetic Interaction Study of Glycopyrrolate and Formoterol in Healthy Volunteers
Acronym: TRIPLE 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CCD-1101-PR-0056; 2011-001552-11 (EudraCT Number)
Record Dates: First submitted 2011-06-09; First posted 2011-07-20 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment R2 (Active Comparator)
  Interventions: Drug: Formoterol
- Treatment R1 (Active Comparator)
  Interventions: Drug: Glycopyrrolate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Treatment T (Experimental)
  Interventions: Drug: Glycopyrrolate + Formoterol

INTERVENTIONS:
Drug: Glycopyrrolate + Formoterol — glycopyrrolate pMDI + formoterol pMDI
  Arms: Treatment T
Drug: Glycopyrrolate — glycopyrrolate pMDI
  Arms: Treatment R1
Drug: Formoterol — formoterol pMDI
  Arms: Treatment R2
Drug: Placebo — placebo pMDI
  Arms: Placebo

SUMMARY:
This study will be carried out in healthy volunteers with the primary objective to evaluate the pharmacokinetic interaction between Glyco and Formoterol administered using a pressurised metered dose inhaler (pMDI).

ELIGIBILITY:
Inclusion Criteria:

* Males and females healthy volunteers aged 18-65 years will be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: formoterol and glyco AUC0-t | from pre-dose to 32 hours after administration
  Area under the plasma concentration curve observed from administration up to the last measurable concentration.
Pharmacokinetics: formoterol and glyco Cmax | from pre-dose to 32 hours after administration
  Maximum plasma concentration

SECONDARY OUTCOMES:
Additional pharmacokinetic variables | from pre-dose to 32 hours post dose
  Plasma Glyco AUC0-30min, AUC0-32h, AUC0-inf, tmax and t1/2 - Plasma Formoterol AUC0-30min, AUC0-24h, AUC0-inf, tmax and t1/2.
Serum potassium | From pre-dose to 24 hours after administration
  Serum potassium Cmin, tmin and AUC0-24h
Plasma glucose | from pre-dose to 24 hours after administration
  Plasma glucose Cmax, tmax and AUC0-24h
Lung function | from pre-dose to 1 hour after administration
  FEV1 in order to assess potential occurrence of paradoxical bronchospasm
Vital signs | from pre-dose to 24 hours after administration
  heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP).
ECG | from pre-dose to 24 hours after administration
  12-lead ECG parameters: HR, RR, PR, QRS, QT, QTcB, QTcF

CONTACTS AND LOCATIONS:
Overall Officials: Lien Gheyle, MD, Principal Investigator — Clinical Pharmacology Unit at SGS Life Sciences - Antwerpen (Belgium)
Locations (1):
- Clinical Pharmacology Unit - SGS Life Science Services, Antwerp, Lange Beeldekensstraat 267, Belgium

REFERENCES:
- See also: CSR Synopsis available in the Chiesi Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-1101-PR-0056.pdf